CLINICAL TRIAL: NCT03517371
Title: Walking and mHealth to Increase Participation in Parkinson Disease
Acronym: WHIPPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Theresa D Ellis, Assistant Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01HD092444 (NIH)
Record Dates: First submitted 2018-04-25; First posted 2018-05-07 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Walking; Exercise; Mobile Health; Physical Therapy; Cognitive Behavioral
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study will take place at Boston University (BU) and Washington University in St. Louis (WU). This is a two-arm, single-blinded, 1-year randomized controlled trial. Persons with mild to moderate PD are randomly assigned to one of two treatment arms. In the mHealth arm, individuals participate in a cognitive-behavioral community-based walking program plus home-based walking enhancing progressive resistance exercises delivered using a mobile health platform. The active control condition receives the same components and dose of walking and exercise but without a cognitive-behavioral approach or the use of mobile health technology.
Who Masked: Outcomes Assessor
Masking Description: Blinded assessors will administer standardizes outcome measures across sites (BU & WU)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth delivered exercise program (Experimental): Participants in the mHealth delivered exercise program have up to 8 in-person visits with a physical therapist over 12 months. The mHealth exercise program, consisting of walking, strengthening and stretching exercises, is prescribed and remotely adapted by a physical therapist over 1 year. Approximately 5-7 exercises are implemented 5 days per week. The exercise program is video-recorded and accessed on a smartphone or computer tablet via an application ("app"). Cognitive-behavioral elements are integrated emphasizing participant engagement in managing their health condition. Components of the mHealth program include goal setting, action planning, automated rewards, self-monitoring of progress and a remote connection to a physical therapist through a messaging feature.
  Interventions: Other: mHealth delivered exercise program
- Exercise only (Active Comparator): Participants in the control group have up to 8 in-person visits with a physical therapist over 12-months - equivalent to the dose provided to the mHealth condition. Participants are instructed by the physical therapist to engage in walking and perform the same progressive resistance and stretching exercises (tailored to their needs and provided in written format) at the same frequency (5x/week) as participants in the mHealth condition. Participants in the control condition are instructed to gradually progress their exercise program and to increase the amount of walking over a 1-year period. No cognitive-behavioral approaches or mHealth technology will be provided.
  Interventions: Other: Exercise only

INTERVENTIONS:
Other: mHealth delivered exercise program — Participants in the mobile health condition have up to 8 in-person visits with a physical therapist over 12 months. The exercise program, consisting of walking, strengthening and stretching exercises, is prescribed through an "app" and remotely adapted by a physical therapist over 1 year. Approximately 5-7 exercises are implemented 5 days per week.
  Arms: mHealth delivered exercise program
Other: Exercise only — Participants in the control group have up to 8 in-person visits with the intervention physical therapist over 12-months. Participants are instructed by the physical therapist to engage in walking and perform progressive resistance and stretching exercises (tailored to their needs and provided in written format) 5 days per week.
  Arms: Exercise only

SUMMARY:
Identifying effective ways to improve function, slow decline and reduce disability is a high priority for people living with Parkinson disease and other chronic conditions. Regular participation in walking is essential to reduce disability and enhance participation in preferred life activities. However, people with chronic conditions are often sedentary, contributing to greater disability. The goal of this work is to determine the benefits of a walking, walking enhancing exercises and cognitive-behavioral strategies delivered using mobile health technology for people with Parkinson disease over a sustained period of time.

DETAILED DESCRIPTION:
Parkinson disease (PD) is one of the most disabling chronic health conditions affecting older adults globally. While advances in medical and surgical management of PD have increased lifespans, these have not effectively altered the progressive decline in physical function and quality of life associated with PD. Identifying effective ways to improve function, slow decline and prevent or reduce disability remains of utmost importance in PD. Of particular concern in PD is gait decline, which is considered a red flag signaling emerging disability. Prior work has shown that people with PD experienced a 12% decline in amount of walking over one year - despite relative stability of motor impairments during that year. Treatment targeting walking, the most rapidly changing aspect of disability in PD, may have the greatest influence on slowing the impact of disease progression on physical function and reducing disability.

Traditionally, rehabilitation has targeted impairments and functional limitations with the expectation that gains would translate into greater participation in real-world activities. However, the evidence suggests that this does not occur. In this proposal, the investigators suggest a paradigm shift in which the primary target of the intervention is real-world walking behavior, as greater walking activity could preserve walking function and slow disability. The primary factors that limit engagement in walking in PD are psychological (e.g., low self-efficacy) rather than physical (e.g., motor impairments) in nature. As such, investigators will evaluate a cognitive-behavioral approach, grounded in social-cognitive theory and targeted at enhancing walking activity. This "connected behavioral approach" links physical therapists to persons with PD using a mobile health (mHealth) platform to deliver strategies to increase self-efficacy and provide goal-oriented, dynamic walking routines and walking enhancing exercises over one year. This approach will be compared to a control intervention which provides equivalent components and dosing of walking and a walking enhancing exercise program delivered by physical therapists but without a cognitive-behavioral mHealth approach. Investigators hypothesize that the mHealth group will demonstrate higher amounts of walking activity and greater walking capacity relative to the control group. With regard to mechanism underlying improvements in the mHealth group, it is hypothesized that self-efficacy will mediate changes in amount of walking and that changes in amount of walking will mediate changes in walking capacity over one year. The insights to be gained regarding mechanisms underlying changes noted will be critical to inform rehabilitation interventions designed to encourage sustained, long-term physical activity. If effective, our "connected behavioral approach" offers a unique, generalizable and scalable means to increase walking activity and improve walking capacity, thereby reducing disability in PD and perhaps in other chronic progressive conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic, typical Parkinson disease according to the UK Brain Bank Criteria;
2. Hoehn & Yahr stages 1-3 (mild to moderate disease severity);
3. Stable on all PD medications for at least 2 weeks prior to study entry;
4. Willing and able to provide informed consent.

Exclusion Criteria:

1. < 18 years of age;
2. Pregnant;
3. diagnosis of atypical Parkinsonism;
4. Hoehn & Yahr stages 4-5
5. a score of > 2 on item 7 of the new freezing of gait questionnaire (moderately or significantly disturbing freezing episodes during daily walking);
6. significant cognitive impairment;
7. unstable medical or concomitant illnesses or psychiatric conditions, which in the opinion of the investigators would preclude successful participation;
8. cardiac problems that interfere with ability to safely exercise
9. orthopedic problems in the lower extremities or spine that may limit walking distance;
10. unable to walk for 10 continuous minutes independently;
11. live in an institution or medical facility (i.e. not in the community)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa D Ellis, PhD, Principal Investigator — Boston University; Gammon M Earhart, PhD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Center for Neurorehabilitation, College of Health & Rehabilitation Sciences, Sargent College, Boston University, Boston, Massachusetts
  - Washington University St. Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shulman LM. Understanding disability in Parkinson's disease. Mov Disord. 2010;25 Suppl 1:S131-5. doi: 10.1002/mds.22789. PMID 20187231
- [Background] Ellis TD, Cavanaugh JT, Earhart GM, Ford MP, Foreman KB, Thackeray A, Thiese MS, Dibble LE. Identifying clinical measures that most accurately reflect the progression of disability in Parkinson disease. Parkinsonism Relat Disord. 2016 Apr;25:65-71. doi: 10.1016/j.parkreldis.2016.02.006. Epub 2016 Feb 2. PMID 26876037
- [Background] Cavanaugh JT, Ellis TD, Earhart GM, Ford MP, Foreman KB, Dibble LE. Capturing ambulatory activity decline in Parkinson's disease. J Neurol Phys Ther. 2012 Jun;36(2):51-7. doi: 10.1097/NPT.0b013e318254ba7a. PMID 22592060
- [Background] Lord S, Godfrey A, Galna B, Mhiripiri D, Burn D, Rochester L. Ambulatory activity in incident Parkinson's: more than meets the eye? J Neurol. 2013 Dec;260(12):2964-72. doi: 10.1007/s00415-013-7037-5. Epub 2013 Jul 31. PMID 23900754
- [Background] Shulman LM, Gruber-Baldini AL, Anderson KE, Vaughan CG, Reich SG, Fishman PS, Weiner WJ. The evolution of disability in Parkinson disease. Mov Disord. 2008 Apr 30;23(6):790-6. doi: 10.1002/mds.21879. PMID 18361474
- [Background] Ellis T, Boudreau JK, DeAngelis TR, Brown LE, Cavanaugh JT, Earhart GM, Ford MP, Foreman KB, Dibble LE. Barriers to exercise in people with Parkinson disease. Phys Ther. 2013 May;93(5):628-36. doi: 10.2522/ptj.20120279. Epub 2013 Jan 3. PMID 23288910
- [Background] Ellis T, Cavanaugh JT, Earhart GM, Ford MP, Foreman KB, Fredman L, Boudreau JK, Dibble LE. Factors associated with exercise behavior in people with Parkinson disease. Phys Ther. 2011 Dec;91(12):1838-48. doi: 10.2522/ptj.20100390. Epub 2011 Oct 14. PMID 22003171
- [Background] Dusseldorp E, van Genugten L, van Buuren S, Verheijden MW, van Empelen P. Combinations of techniques that effectively change health behavior: evidence from Meta-CART analysis. Health Psychol. 2014 Dec;33(12):1530-40. doi: 10.1037/hea0000018. Epub 2013 Nov 25. PMID 24274802
- [Background] Whitehead L, Seaton P. The Effectiveness of Self-Management Mobile Phone and Tablet Apps in Long-term Condition Management: A Systematic Review. J Med Internet Res. 2016 May 16;18(5):e97. doi: 10.2196/jmir.4883. PMID 27185295
- [Background] Tudor-Locke C, Bassett DR Jr. How many steps/day are enough? Preliminary pedometer indices for public health. Sports Med. 2004;34(1):1-8. doi: 10.2165/00007256-200434010-00001. PMID 14715035
- [Background] Dontje ML, de Greef MH, Speelman AD, van Nimwegen M, Krijnen WP, Stolk RP, Kamsma YP, Bloem BR, Munneke M, van der Schans CP. Quantifying daily physical activity and determinants in sedentary patients with Parkinson's disease. Parkinsonism Relat Disord. 2013 Oct;19(10):878-82. doi: 10.1016/j.parkreldis.2013.05.014. Epub 2013 Jun 12. PMID 23769178
- [Background] Oguh O, Eisenstein A, Kwasny M, Simuni T. Back to the basics: regular exercise matters in parkinson's disease: results from the National Parkinson Foundation QII registry study. Parkinsonism Relat Disord. 2014 Nov;20(11):1221-5. doi: 10.1016/j.parkreldis.2014.09.008. Epub 2014 Sep 16. PMID 25258329
- [Background] Corcos DM, Robichaud JA, David FJ, Leurgans SE, Vaillancourt DE, Poon C, Rafferty MR, Kohrt WM, Comella CL. A two-year randomized controlled trial of progressive resistance exercise for Parkinson's disease. Mov Disord. 2013 Aug;28(9):1230-40. doi: 10.1002/mds.25380. Epub 2013 Mar 27. PMID 23536417
- [Background] LaHue SC, Comella CL, Tanner CM. The best medicine? The influence of physical activity and inactivity on Parkinson's disease. Mov Disord. 2016 Oct;31(10):1444-1454. doi: 10.1002/mds.26728. PMID 27477046
- [Background] Petzinger GM, Fisher BE, McEwen S, Beeler JA, Walsh JP, Jakowec MW. Exercise-enhanced neuroplasticity targeting motor and cognitive circuitry in Parkinson's disease. Lancet Neurol. 2013 Jul;12(7):716-26. doi: 10.1016/S1474-4422(13)70123-6. PMID 23769598
- [Background] Hirsch MA, Iyer SS, Sanjak M. Exercise-induced neuroplasticity in human Parkinson's disease: What is the evidence telling us? Parkinsonism Relat Disord. 2016 Jan;22 Suppl 1:S78-81. doi: 10.1016/j.parkreldis.2015.09.030. Epub 2015 Sep 15. PMID 26439945
- [Background] Uc EY, Doerschug KC, Magnotta V, Dawson JD, Thomsen TR, Kline JN, Rizzo M, Newman SR, Mehta S, Grabowski TJ, Bruss J, Blanchette DR, Anderson SW, Voss MW, Kramer AF, Darling WG. Phase I/II randomized trial of aerobic exercise in Parkinson disease in a community setting. Neurology. 2014 Jul 29;83(5):413-25. doi: 10.1212/WNL.0000000000000644. Epub 2014 Jul 2. PMID 24991037
- [Background] Shulman LM, Katzel LI, Ivey FM, Sorkin JD, Favors K, Anderson KE, Smith BA, Reich SG, Weiner WJ, Macko RF. Randomized clinical trial of 3 types of physical exercise for patients with Parkinson disease. JAMA Neurol. 2013 Feb;70(2):183-90. doi: 10.1001/jamaneurol.2013.646. PMID 23128427
- [Background] Williams SL, French DP. What are the most effective intervention techniques for changing physical activity self-efficacy and physical activity behaviour--and are they the same? Health Educ Res. 2011 Apr;26(2):308-22. doi: 10.1093/her/cyr005. Epub 2011 Feb 14. PMID 21321008
- [Background] Richardson J, Loyola-Sanchez A, Sinclair S, Harris J, Letts L, MacIntyre NJ, Wilkins S, Burgos-Martinez G, Wishart L, McBay C, Martin Ginis K. Self-management interventions for chronic disease: a systematic scoping review. Clin Rehabil. 2014 Nov;28(11):1067-77. doi: 10.1177/0269215514532478. Epub 2014 Apr 30. PMID 24784031
- [Background] Archer KR, Devin CJ, Vanston SW, Koyama T, Phillips SE, Mathis SL, George SZ, McGirt MJ, Spengler DM, Aaronson OS, Cheng JS, Wegener ST. Cognitive-Behavioral-Based Physical Therapy for Patients With Chronic Pain Undergoing Lumbar Spine Surgery: A Randomized Controlled Trial. J Pain. 2016 Jan;17(1):76-89. doi: 10.1016/j.jpain.2015.09.013. Epub 2015 Oct 23. PMID 26476267
- [Background] Vassilev I, Rowsell A, Pope C, Kennedy A, O'Cathain A, Salisbury C, Rogers A. Assessing the implementability of telehealth interventions for self-management support: a realist review. Implement Sci. 2015 Apr 24;10:59. doi: 10.1186/s13012-015-0238-9. PMID 25906822
- [Background] Hamine S, Gerth-Guyette E, Faulx D, Green BB, Ginsburg AS. Impact of mHealth chronic disease management on treatment adherence and patient outcomes: a systematic review. J Med Internet Res. 2015 Feb 24;17(2):e52. doi: 10.2196/jmir.3951. PMID 25803266
- [Background] Moller AC, Merchant G, Conroy DE, West R, Hekler E, Kugler KC, Michie S. Applying and advancing behavior change theories and techniques in the context of a digital health revolution: proposals for more effectively realizing untapped potential. J Behav Med. 2017 Feb;40(1):85-98. doi: 10.1007/s10865-016-9818-7. Epub 2017 Jan 5. PMID 28058516
- [Background] Geuens J, Swinnen TW, Westhovens R, de Vlam K, Geurts L, Vanden Abeele V. A Review of Persuasive Principles in Mobile Apps for Chronic Arthritis Patients: Opportunities for Improvement. JMIR Mhealth Uhealth. 2016 Oct 13;4(4):e118. doi: 10.2196/mhealth.6286. PMID 27742604
- [Background] Lee AC, Harada N. Telehealth as a means of health care delivery for physical therapist practice. Phys Ther. 2012 Mar;92(3):463-8. doi: 10.2522/ptj.20110100. Epub 2011 Dec 1. No abstract available. PMID 22135703
- [Background] Cavanaugh JT, Ellis TD, Earhart GM, Ford MP, Foreman KB, Dibble LE. Toward Understanding Ambulatory Activity Decline in Parkinson Disease. Phys Ther. 2015 Aug;95(8):1142-50. doi: 10.2522/ptj.20140498. Epub 2015 Apr 9. PMID 25858971
- [Background] Motl RW, Pilutti LA, Learmonth YC, Goldman MD, Brown T. Clinical importance of steps taken per day among persons with multiple sclerosis. PLoS One. 2013 Sep 4;8(9):e73247. doi: 10.1371/journal.pone.0073247. eCollection 2013. PMID 24023843
- [Background] Speelman AD, van Nimwegen M, Borm GF, Bloem BR, Munneke M. Monitoring of walking in Parkinson's disease: validation of an ambulatory activity monitor. Parkinsonism Relat Disord. 2011 Jun;17(5):402-4. doi: 10.1016/j.parkreldis.2011.02.006. Epub 2011 Mar 1. No abstract available. PMID 21367643
- [Background] Tudor-Locke C, Leonardi C, Johnson WD, Katzmarzyk PT, Church TS. Accelerometer steps/day translation of moderate-to-vigorous activity. Prev Med. 2011 Jul-Aug;53(1-2):31-3. doi: 10.1016/j.ypmed.2011.01.014. Epub 2011 Feb 2. PMID 21295063
- [Background] van Nimwegen M, Speelman AD, Overeem S, van de Warrenburg BP, Smulders K, Dontje ML, Borm GF, Backx FJ, Bloem BR, Munneke M; ParkFit Study Group. Promotion of physical activity and fitness in sedentary patients with Parkinson's disease: randomised controlled trial. BMJ. 2013 Mar 1;346:f576. doi: 10.1136/bmj.f576. PMID 23457213
- [Background] Ellis T, Latham NK, DeAngelis TR, Thomas CA, Saint-Hilaire M, Bickmore TW. Feasibility of a virtual exercise coach to promote walking in community-dwelling persons with Parkinson disease. Am J Phys Med Rehabil. 2013 Jun;92(6):472-81; quiz 482-5. doi: 10.1097/PHM.0b013e31828cd466. PMID 23552335
- [Background] Tudor-Locke C. Walk more (frequently, farther, faster): the perfect preventive medicine. Prev Med. 2012 Dec;55(6):540-1. doi: 10.1016/j.ypmed.2012.07.009. Epub 2012 Jul 20. No abstract available. PMID 22819847
- [Derived] Paul SS, Porciuncula F, Cavanaugh JT, Rawson KS, Nordahl TJ, Baker TC, Duncan RP, Earhart GM, Ellis TD. Causal Mediation Analysis of Factors Influencing Physical Activity and Community Access Among People With Mild-to-Moderate Parkinson Disease. Arch Phys Med Rehabil. 2025 Jun;106(6):871-879. doi: 10.1016/j.apmr.2024.10.012. Epub 2024 Nov 5. PMID 39505247
- [Derived] Girnis JL, Cavanaugh JT, Baker TC, Duncan RP, Fulford D, LaValley MP, Lawrence M, Nordahl T, Porciuncula F, Rawson KS, Saint-Hilaire M, Thomas CA, Zajac JA, Earhart GM, Ellis TD. Natural Walking Intensity in Persons With Parkinson Disease. J Neurol Phys Ther. 2023 Jul 1;47(3):146-154. doi: 10.1097/NPT.0000000000000440. Epub 2023 Apr 4. PMID 37016469
- [Derived] Zajac JA, Cavanaugh JT, Baker T, Colon-Semenza C, DeAngelis TR, Duncan RP, Fulford D, LaValley M, Nordahl T, Rawson KS, Saint-Hilaire M, Thomas CA, Earhart GM, Ellis TD. Are Mobile Persons With Parkinson Disease Necessarily More Active? J Neurol Phys Ther. 2021 Oct 1;45(4):259-265. doi: 10.1097/NPT.0000000000000362. PMID 34091569
- [Derived] Rawson KS, Cavanaugh JT, Colon-Semenza C, DeAngelis T, Duncan RP, Fulford D, LaValley MP, Mazzoni P, Nordahl T, Quintiliani LM, Saint-Hilaire M, Thomas CA, Earhart GM, Ellis TD. Design of the WHIP-PD study: a phase II, twelve-month, dual-site, randomized controlled trial evaluating the effects of a cognitive-behavioral approach for promoting enhanced walking activity using mobile health technology in people with Parkinson-disease. BMC Neurol. 2020 Apr 20;20(1):146. doi: 10.1186/s12883-020-01718-z. PMID 32312243

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in February 2019 and concluded in March 2023. We experienced pauses in recruiting new participants during COVID 2020-2021. For already enrolled participants, we continued collection of measures that could be done remotely. Recruitment was via flyers which were available at physical therapy clinics, movement disorder clinics, support groups, and health fairs and events.
Pre-assignment Details: Participants were excluded during in-person screening if they had significant cognitive impairment (Mini-Mental Status Examination < 24), disturbing freezing of gait episodes during daily walking (score of ≥ 2 on item 7 of New Freezing of Gait Questionnaire, resting tachycardia (>120 beats/min), uncontrolled BP (resting systolic BP>180 mmHg or diastolic BP>100 mmHg)), unstable medical illnesses or conditions that would preclude successful participation, and/or Modified Hoehn & Yahr stage >3.
Period: Overall Study
Arm/Group | mHealth Delivered Exercise Program | Exercise Only
Started | 73 | 67
Completed | 58 | 48
Not Completed | 15 | 19
Not completed — Adverse Event | 8 | 9
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Not idiopathic Parkinson's disease | 0 | 3
Not completed — COVID restrictions | 2 | 0
Not completed — Receiving DBS Surgery | 0 | 1

BASELINE CHARACTERISTICS:
Population: No difference.
Groups:
- Total: Total of all reporting groups
Arm/Group | mHealth Delivered Exercise Program | Exercise Only | Total
Number analyzed (Participants) | 73 | 67 | 140
Age, Continuous [Mean (Standard Deviation); unit: age, continuous, in years] — Age, continuous, in years
  age, continuous, in years | 68.25 (8.37) | 67.21 (7.79) | 67.75 (8.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 32 | 65
  Male | 40 | 35 | 75
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 69 | 63 | 132
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 71 | 67 | 138
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Walking Activity
Description: Change in the average number of steps walked per day over the one year study. Participants wore the step watch for one week before starting the program as part of their baseline visit and one week at the end of the year program as part of their 12-month visit. Daily steps were averaged at baseline and 12-month and a change score was computed (average of daily steps at 12-Months minus average of daily steps at baseline).
Time Frame: 12 months
Population: There were 15 participants who withdrew in mHealth group and 19 participant who withdrew in the exercise group. In addition, one participant was missing daily step data at random at 12 months in mHealth, and one participant was missing data due to a technical issue with the step watch in the exercise group.
Measure: Mean (Standard Deviation); unit: change in average daily steps
Arm/Group | mHealth Delivered Exercise Program | Exercise Only
Number analyzed (Participants) | 57 | 47
change in average daily steps | -207.59 (2749.39) | -135.24 (2403.17)
Statistical Analysis 1: Comparison: mHealth Delivered Exercise Program vs Exercise Only; Test type: Superiority; p = .89, t-test, 2 sided; Mean Difference (Final Values) = 72.35, 95% CI 2-sided [-943.34 to 1088.04]

2. Primary Outcome: Walking Intensity
Description: Change in the average number of moderate intensity minutes over the one year study. Moderate intensity minutes is defined as the number of minutes in which >100 steps were accumulated. Participants wore the step watch for one week before starting the program as part of their baseline visit and one week at the end of the year program as part of their 12-month visit. Moderate intensity minutes were averaged at baseline and 12-month and a change score was computed (average of moderate intensity minutes at 12-Months minus average of moderate intensity minutes at baseline).
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change in average moderate intensity min
Arm/Group | mHealth Delivered Exercise Program | Exercise Only
Number analyzed (Participants) | 57 | 47
change in average moderate intensity min | 1.67 (9.41) | 1.33 (8.07)
Statistical Analysis 1: Comparison: mHealth Delivered Exercise Program vs Exercise Only; Test type: Superiority; p = .42, t-test, 2 sided; Mean Difference (Final Values) = -.35, 95% CI 2-sided [-3.80 to 3.10]

3. Secondary Outcome: Walking Capacity - Six Minute Walk Distance
Description: Change in the number of meters walked during the six-minute walk test over the one year study. The distance in meters is reported. Participants completed the six-minute walk before starting the program as part of their baseline visit and at the end of the year program as part of their 12-month visit. A change score was computed - the number of meters walked at 12 months minus the number of meters walked at baseline).
Time Frame: 12 months
Population: There were 15 participants who withdrew in the mHealth group and 19 participants who withdrew in the exercise group. Due to COVID restrictions, we were unable to complete measures that required participants to come in-person, thus we are missing data on this measure for 17 more people in the mHealth group and 19 more people in the exercise group. In addition, one participant in mHealth and one participant in exercise group did not complete this measure at 12-month due to physical reasons.
Measure: Mean (Standard Deviation); unit: change in meters walked
Arm/Group | mHealth Delivered Exercise Program | Exercise Only
Number analyzed (Participants) | 40 | 28
change in meters walked | 15.63 (57.02) | 17.79 (37.12)
Statistical Analysis 1: Comparison: mHealth Delivered Exercise Program vs Exercise Only; Test type: Superiority; p = .85, t-test, 2 sided; Levene's test significant, equal variances not assumed values reported; Median Difference (Final Values) = 2.17, 95% CI 2-sided [-20.64 to 24.97]

4. Secondary Outcome: Walking Capacity - Ten Meter Walk Test
Description: Change in the number of meters per second walked during the ten-meter walk test (comfortable forward pace) over the one year study. The distance in meters per second are reported. Participants completed the ten-meter walk test before starting the program as part of their baseline visit and at the end of the year program as part of their 12-month visit. A change score was computed - the number of meters per second walked at 12-months minus the number of meters per second walked at baseline).
Time Frame: 12 months
Population: There were 15 participants who withdrew in the mHealth group and 19 participants who withdrew in the exercise group. Due to COVID restrictions, we were unable to complete measures that required participants to come in-person, thus we are missing data on this measure for 17 more people in the mHealth group and 19 more people in the exercise group. In addition, one participant in mHealth did not complete this measure at 12 months due to physical reasons.
Measure: Mean (Standard Deviation); unit: change in meters per second
Arm/Group | mHealth Delivered Exercise Program | Exercise Only
Number analyzed (Participants) | 40 | 29
change in meters per second | .027 (.146) | .019 (.154)
Statistical Analysis 1: Comparison: mHealth Delivered Exercise Program vs Exercise Only; Test type: Superiority; p = .824, t-test, 2 sided; Mean Difference (Final Values) = -.008, 95% CI 2-sided [-.081 to .065]

ADVERSE EVENTS:
Time Frame: Information about adverse events were collected from active participants - either until they withdrew or completed the one-year study.
Arm/Group | mHealth Delivered Exercise Program | Exercise Only
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/67
Serious Adverse Events (participants affected / at risk) | 15/73 | 17/67
Other Adverse Events (participants affected / at risk) | 39/73 | 35/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mHealth Delivered Exercise Program (N=73) | Exercise Only (N=67)
Retinal Detachment (Eye disorders) | 0 (0) | 1 (1)
Esophageal Spasm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gait Disturbance (General disorders) | 0 (0) | 1 (1)
Gallbladder Pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 8 (8)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Renal Calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Cognitive Disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Neoplasm - Salivary Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm - Ovarian (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Device Related Infection (Infections and infestations) | 1 (1) | 0 (0)
Lower Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Myocardial Infection (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mHealth Delivered Exercise Program (N=73) | Exercise Only (N=67)
Fall (Injury, poisoning and procedural complications) | 15 (19) | 14 (17)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (7)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 19 (24) | 14 (18)

LIMITATIONS AND CAVEATS:
Limitations included slower than expected recruitment levels and higher levels of attrition than projected due to COVID-19 restrictions. To comply with University and Governmental guidelines, in-person visits were put on hold for several months in 2020 and 2021. This prevented collection of secondary outcomes (6-minute and 10 meter walks). However, we were able to continue collection of the primary outcomes (daily steps, moderate intensity minutes) via the step watch remotely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT03517371/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT03517371/SAP_001.pdf
  • Informed Consent Form (2022-05-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT03517371/ICF_002.pdf